CLINICAL TRIAL: NCT00572715
Title: Acute Kidney Injury in Neonates
Status: Withdrawn | Type: Observational
Why Stopped: Investigator's decision:Did not open to enrollment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Askenazi, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: X070927001
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Acute Kidney Injury
Keywords: kidney; neonates
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Inclusion criteria - Families of infants (birthweight >1500g) be asked to participate in the study.
  Exclusion criteria - Infants with prenatal renal ultrasound diagnosis of severe hydronephrosis or other known renal abnormalities will be excluded

SUMMARY:
Our first aim is to describe how common a sudden decrease in renal function happens in infants in a neonatal intensive care unit. We also want to see how a sudden loss of renal function affects survival. Finally, we will explore non-invasive markers to identify a sudden decrease in renal function from urinary samples.

DETAILED DESCRIPTION:
Advancements in the field of peri-natal medicine has improved the survival of critically ill neonates but yet many still do not survive, and many more are left with long-term damage to vital organ systems. Very little data is available on the impact that acute kidney injury (AKI) has on survival in term neonates, but adult and pediatric studies that show that even mild AKI independently impacts survival after correcting for severity of illness. The role that AKI impacts survival in neonates is likely to be greater than adults as this acute injury occurs in context of impaired and ongoing kidney development.

Our ability to improve outcomes in children and adults with AKI has been hampered by the inability to recognize AKI early in the disease process. Thus, the work on early non-invasive biomarkers of renal injury has brought great optimism to the field of AKI. Serum and urinary levels of neutrophil gelatinase-associated lipocalin (NGAL), urinary interleukin 18 (IL-18) others are markedly elevated several hours after AKI as opposed to serum creatinine which takes days to rise after the inciting event. Early non-invasive biomarkers of AKI have not been tested in neonates.

Inclusion criteria - Families of infants (birthweight >1500g) be asked to participate in the study.

Exclusion criteria - Infants with prenatal renal ultrasound diagnosis of severe hydronephrosis or other known renal abnormalities will be excluded

ELIGIBILITY:
Inclusion Criteria:

* Families of infants (birthweight >1500g) be asked to participate in the study.

Exclusion Criteria:

* Infants with prenatal renal ultrasound diagnosis of severe hydronephrosis or other known renal abnormalities will be excluded

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion criteria - Families of infants (birthweight >1500g) be asked to participate in the study.
  Exclusion criteria - Infants with prenatal renal ultrasound diagnosis of severe hydronephrosis or other known renal abnormalities will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01-31; Study Completion 2010-01-31 (Actual)

PRIMARY OUTCOMES:
Characterize the incidence and risk factors of AKI in critically ill neonates | 2 years

SECONDARY OUTCOMES:
Compare Hospital outcomes of critically ill neonates with and without AKI. Test the ability of known noninvasive urinary biomarkers ability to detect AKI in neonates | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States